CLINICAL TRIAL: NCT06751797
Title: Balance Confidence, Kinesiophobia, and Associated Factors in Parkinson's Disease: A Controlled Study
Brief Title: Balance Confidence and Kinesiophobia in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH13
Record Dates: First submitted 2024-12-09; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease group: Patient with parkinson disease
  Interventions: Other: No intervention
- Control group: Healthy controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
31 patients aged 50-80 years diagnosed with idiopathic Parkinson's disease (Modified Hoehn-Yahr stages 1-3) and 31 healthy volunteers. At the start of the study, sociodemographic data for all participants will be recorded. To assess the mental and functional status of Parkinson's disease patients, the Mini-Mental State Examination (MMSE) and the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) will be used. Balance confidence levels will be assessed using the Activities-specific Balance Confidence Scale-6 (ABC-6), overall balance using the Berg Balance Scale (BBS), fear of falling using the Falls Efficacy Scale (FES), and kinesiophobia levels using the Tampa Scale of Kinesiophobia (TSK).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Parkinson's Disease by a neurology specialist.
* Modified Hoehn-Yahr Staging Scale classification between stages 1-3.
* Mini-Mental State Examination (MMSE) score of 24 or higher.
* Age between 50-80 years.
* Volunteered to participate in the study.

Exclusion Criteria:

* Use of medications, apart from routine Parkinson's disease treatments, that could affect balance or muscle strength.
* Presence of neurological or musculoskeletal conditions other than Parkinson's disease.
* Refusal to participate in the study.
* Presence of psychiatric disorders.
* Presence of cognitive impairments.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinson disease and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Balance Confidence (ABC-6 Scale) | Baseline
  Evaluated using the Activities-specific Balance Confidence Scale-6 (ABC-6), which measures participants' confidence in maintaining balance during various daily activities. Lower scores indicate reduced balance confidence, a common issue in Parkinson's disease.
  In the ABC-6 scale, the minimum score is 0% (no confidence), the maximum score is 100% (full confidence), and the total score is calculated as the average of the percentages given for all activities.

SECONDARY OUTCOMES:
Balance Level (Berg Balance Scale) | Baseline
  Assessed using the Berg Balance Scale (BBS) to quantify participants' overall balance performance through functional balance tasks. Lower scores reflect greater balance impairment. In the Berg Balance Scale (BBS), the minimum score is 0 (indicating poor balance), and the maximum score is 56 (indicating excellent balance). The total score is the sum of the individual scores from 14 items, each rated on a 5-point scale (0-4).
Fear of Falling (Falls Efficacy Scale) | Baseline
  Measured using the Falls Efficacy Scale (FES), which evaluates fear of falling during specific activities. Higher scores indicate a greater fear of falling, often linked to reduced mobility and participation.
  In the Falls Efficacy Scale (FES), the minimum score is 10 (indicating no fear of falling), and the maximum score is 100 (indicating extreme fear of falling). The score is calculated by summing the ratings for 10 items, each scored on a 1-10 scale.
Kinesiophobia (Tampa Scale of Kinesiophobia) | Baseline
  Assessed with the Tampa Scale of Kinesiophobia (TSK) to measure fear of movement or re-injury. Higher scores indicate greater kinesiophobia, potentially limiting physical activity in Parkinson's patients.
  In the Tampa Scale of Kinesiophobia (TSK), the minimum score is 17 (indicating low kinesiophobia), and the maximum score is 68 (indicating high kinesiophobia). The total score is obtained by summing the ratings for 17 items, each scored on a 1-4 scale.
Mental Status (MMSE) | Baseline
  The Mini-Mental State Examination (MMSE) evaluates cognitive function, including orientation, memory, attention, language, and visuospatial skills, with scores ranging from 0 (severe cognitive impairment) to 30 (normal cognitive function).
Functional status (MDS-UPDRS) | Baseline
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assesses functional status and disease severity in Parkinson's disease, encompassing non-motor and motor experiences of daily living, motor examination, and motor complications. The total score ranges from 0 (no symptoms) to 260 (severe symptoms), with higher scores indicating greater disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No